CLINICAL TRIAL: NCT02228980
Title: Immunogenicity and Safety of a Single Dose (Subjects From 3 Years of Age) or Two Doses Given 28 Days Apart (Children From 6 to 35 Months of Age) of a Trivalent Inactivated Influenza Vaccine Produced at Shenzhen, China
Brief Title: Study of a Single Dose or Two Doses of a Trivalent Inactivated Influenza Vaccine Produced at Shenzhen, China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FST01; U1111-1143-8684 (Other: WHO); CTR20140452 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: Influenza; Trivalent influenza vaccine; Sanofi Pasteur Shenzhen trivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects aged 6 to 35 months (Group 1) (Experimental): Participants aged 6 months to 35 months will receive two 0.25 mL doses of SP Shz TIV given 28 days apart.
  Interventions: Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation
- Subjects aged 3 to 17 years (Group 2) (Experimental): Participants aged 3 years to 17 years will receive a single 0.5 mL dose of SP Shz TIV
  Interventions: Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation
- Subjects aged 18 to 60 years (Group 3) (Experimental): Participants aged 18 years to 60 years will receive a single 0.5 mL dose of SP Shz TIV
  Interventions: Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation
- Subjects aged 61 years or older (Group 4) (Experimental): Participants aged 61 years or older will receive a single 0.5 mL dose of SP Shz TIV
  Interventions: Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation

INTERVENTIONS:
Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation — 0.25 mL Intramuscular (2 doses given 28 days apart)
  Arms: Subjects aged 6 to 35 months (Group 1)
Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation — 0.5 mL Intramuscular
  Arms: Subjects aged 3 to 17 years (Group 2)
Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation — 0.5 mL Intramuscular
  Arms: Subjects aged 18 to 60 years (Group 3)
Biological: Shenzhen trivalent influenza vaccine (split virion, inactivated) North Hemisphere (NH) formulation — 0.5 mL Intramuscular
  Arms: Subjects aged 61 years or older (Group 4)

SUMMARY:
The main purpose of this trial is to describe the product profile in terms of immunogenicity and safety following administration of trivalent influenza vaccine (split-virion, inactivated) produced at Shenzhen (SP Shz TIV).

Primary objective:

* To describe in each group the immune response induced by a single dose (subjects aged ≥ 3 years) or by two doses (subjects aged 6 to 35 months) of SP Shz-TIV.

Secondary objective:

* To describe in each group the safety profile of the vaccine after a single dose (subjects aged ≥ 3 years) or after each and any dose administered (subjects aged 6-35 months).

DETAILED DESCRIPTION:
Healthy subjects will be included to receive one or two doses of SP Shz TIV The study will assess the immunogenicity and safety of a single dose (in subjects from 3 years) or two doses of SP Shz TIV vaccine given 28 days apart (pediatric population from 6 to 35 months).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 6 months on the day of inclusion
* Informed Consent Form has been signed and dated:

  * by the parent(s) or legally acceptable representative, if applicable, for subjects <18 years of age. Additionally, an assent form has been signed by the subject if aged 10 to 17 years (based on local regulations).
  * by the subject himself/herself for subjects ≥18 years of age.
* Subject and parent(s)/legally acceptable representative (if applicable) are able to attend all scheduled visits and to comply with all trial procedures
* For subjects aged 6-35 months only: Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg
* For subjects aged 3-8 years only: Subject has previously received at least one dose of influenza vaccine in the past years or has a history of prior exposure to influenza virus through natural infection.

Exclusion Criteria:

* Subject is pregnant (positive urine pregnancy test), or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine or planned receipt of any vaccine within the period from 2 weeks before to 2 weeks after trial vaccination (subjects aged ≥3 years) or within the period from 2 weeks before the first trial vaccination to 2 weeks after the second trial vaccination (subjects aged 6-35 months)
* For subjects aged 6-35 months only: Previous vaccination against influenza (i.e. 2 consecutive doses of influenza vaccine [same seasonal strain composition]) any time prior to study enrollment or history of prior exposure to influenza virus through natural infection
* Vaccination against influenza given in the past 6 months with any influenza vaccine or planned receipt of influenza vaccination during the present study
* Receipt of immune globulins, blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Reported history of seropositivity for Human Immunodeficiency Virus (HIV), after questioning the subject or the subject's parents or another legally acceptable representative
* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substance
* Self-reported thrombocytopenia, as reported by the subject, parent or legally acceptable representative contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination upon investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Nanning, Guangxi, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 05 September 2014 to 09 October 2014 at 1 clinical center at the Province of Guangxi China.
Pre-assignment Details: A total of 602 participants who met all of the inclusion and none of the exclusion criteria were vaccinated in this study.
Groups:
- Age 6 to 35 Months Group: Participants 6 to 35 months of age received two 0.25 mL doses of trivalent influenza vaccine (split-virion, inactivated) given 28 days apart.
- Age 3 to 17 Years Group: Participants 3 to 17 years of age received a single 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Age 18 to 60 Years Group: Participants 18 to 60 years of age received a single 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Age ≥61 Years Group: Participants ≥61 years of age received a single 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
Period: Overall Study
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 18 to 60 Years Group | Age ≥61 Years Group
Started | 150 | 150 | 151 | 151
Completed | 126 | 147 | 149 | 148
Not Completed | 24 | 3 | 2 | 3
Not completed — Adverse Event | 14 | 0 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 18 to 60 Years Group | Age ≥61 Years Group | Total
Number analyzed (Participants) | 150 | 150 | 151 | 151 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 150 | 150 | 0 | 0 | 300
  Between 18 and 65 years | 0 | 0 | 151 | 41 | 192
  >=65 years | 0 | 0 | 0 | 110 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.45 (0.597) | 8.55 (3.09) | 46.5 (11.2) | 69.8 (6.37) | 31.5 (5.31425)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 70 | 114 | 79 | 331
  Male | 82 | 80 | 37 | 72 | 271
Region of Enrollment [Number; unit: Participants]
  China | 150 | 150 | 151 | 151 | 602

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Influenza Antibodies Before and Following Vaccination With a Trivalent Inactivated Influenza Vaccine
Description: Anti-hemagglutinin (HA) antibody titers were measured using the Hemagglutination Inhibition (HAI) technique.
Time Frame: Day 0 (pre-vaccination) up to Day 28 or Day 56 (Age 6 to 35 Months Group) post-vaccination
Population: Geometric mean titers against the trivalent inactivated influenza vaccine antigens were assessed in the Immunogenicity Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Groups:
- Age 3 to 17 Years Group: Participants 3 to 17 years of age received a single 0.5-mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Age 8 to 60 Years Group: Participants 18 to 60 years of age received a single 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 8 to 60 Years Group | Age ≥61 Years Group
Number analyzed (Participants) | 150 | 150 | 151 | 151
Titers (1/dilution)
  A/H1N1 (Pre-dose; N=150,150,151,151) | 12.8 [10.5 to 15.6] | 24.3 [20.1 to 29.4] | 11.2 [9.49 to 13.1] | 9 [7.68 to 10.5]
  A/H1N1 (Post-dose; N=125,145,149,145) | 152.2 [120 to 193] | 300.7 [243 to 372] | 188.3 [158 to 224] | 144 [116 to 180]
  A/H3N2 (Pre-dose; n=150,150,151,151) | 14.3 [11.3 to 18.1] | 62 [51.5 to 74.8] | 12.2 [10.4 to 14.4] | 21.1 [16.9 to 26.5]
  A/H3N2 (Post-dose; N=125,146,149,147) | 235.9 [191 to 291] | 236.2 [207 to 270] | 166.1 [140 to 197] | 237.8 [198 to 285]
  B (Pre-dose; N=150,150,151,151) | 5.9 [5.49 to 6.30] | 17.7 [15.0 to 20.9] | 16.3 [13.7 to 19.5] | 15.3 [12.8 to 18.2]
  B (Post-dose; N=123,146,149,148) | 108.5 [90.9 to 129] | 216.8 [180 to 261] | 202.8 [168 to 245] | 170 [140 to 207]

2. Other Pre Specified Outcome: Percentage of Participants With Seroprotection Before and Following Vaccination With a Trivalent Inactivated Influenza Vaccine
Description: Anti-hemagglutinin (HA) antibody titers were measured using the Hemagglutination Inhibition (HAI) technique. Seroprotection was defined as titers ≥ 40 (1/dil) on Day 0 and Day 28 or Day 56.
Time Frame: Day 0 (pre-vaccination) up to Day 28 or Day 56 (Age 6 to 35 Months Group) post-vaccination
Population: Seroprotection against the trivalent inactivated influenza vaccine were assessed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 8 to 60 Years Group | Age ≥61 Years Group
Number analyzed (Participants) | 150 | 150 | 151 | 151
Percentage of participants
  A/H1N1 (Pre-dose; N=150,150,151,151) | 31.3 | 45.3 | 17.2 | 14.6
  A/H1N1 (Post-dose; N=125,145,149,145) | 88.8 | 94.5 | 96.6 | 89.7
  A/H3N2 (Pre-dose; N=150,150,151,151) | 32.0 | 78.0 | 21.9 | 39.1
  A/H3N2 (Post-dose; N=125,146,149,147) | 98.4 | 99.3 | 95.3 | 95.9
  B (Pre-dose; N=150,150,151,151) | 1.3 | 30.0 | 29.8 | 23.8
  B (Post-dose; N=123,146,149,148) | 93.5 | 95.2 | 98.7 | 93.9

3. Other Pre Specified Outcome: Percentage of Participants With Seroconversion or Significant Increase in Influenza Antibody Titers Following Vaccination With a Trivalent Inactivated Influenza Vaccine
Description: Anti hemagglutinin (HA) antibody titers were measured using the Hemagglutination Inhibition (HAI) technique. Seroconversion was defined as titers < 10 (1/dil) on Day 0 and post vaccination titer ≥ 40 (1/dil) on Day 28 or Day 56 or significant increase was titers ≥ 10 (1/dil) on Day 0 and ≥ 4-fold increase of post-vaccination titer on Day 28 or Day 56.
Time Frame: Day 0 (pre-vaccination) up to Day 28 or Day 56 (Age 6 to 35 Months Group) post-vaccination
Population: Seroconversion or significant increase against the trivalent inactivated influenza vaccine were assessed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Age 3 to 17 Years Group: Participants 3 to 17 years of age received a 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Age 18 to 60 Years Group: Participants 18 to 60 years of age received a 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Age ≥61 Years Group: Participants ≥61 years of age received a 0.5 mL dose of trivalent influenza vaccine (split-virion, inactivated).
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 18 to 60 Years Group | Age ≥61 Years Group
Number analyzed (Participants) | 125 | 146 | 149 | 148
Percentage of participants
  A/H1N1 (N=125,145,149,145) | 86.4 | 79.3 | 91.3 | 84.1
  A/H3N2 (N=125,146,149,147) | 90.4 | 56.2 | 83.2 | 78.2
  B (N=123,146,149,148) | 93.5 | 82.2 | 85.9 | 80.4

4. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions Following Vaccination With a Trivalent Inactivated Influenza Vaccine
Description: Solicited injection site: Tenderness/Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited Systemic: Fever, (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability (≤ 23 months); Fever, Headache, Malaise, Myalgia, and Shivering (≥2 years).
  Grade 3: Tenderness - Cries if injected limb is moved; Pain - Incapacitating; Erythema, Swelling, Induration, Ecchymosis, ≥ 50 mm or 100 mm age ≥ 12 years: Fever >39.5˚C; Crying abnormal - >3 hours; Drowsiness - Difficulty waking; Appetite lost - Refuses ≥3 meals; Irritability - Inconsolable; Vomiting - ≥6 incidents per 24 hours: Fever ≥39.0˚C; Headache, Malaise, Myalgia, and Shivering - Prevents activity (≥ 2 years)
Time Frame: Day 0 up to Day 7 post any vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Population.
Measure: Number; unit: Participants
Arm/Group | Age 6 to 35 Months Group | Age 3 to 17 Years Group | Age 18 to 60 Years Group | Age ≥61 Years Group
Number analyzed (Participants) | 150 | 150 | 151 | 151
Participants
  Injection site Tenderness/Pain (N=140,148,150,151) | 38 | 52 | 25 | 12
  Grade 3 Tenderness/Pain (N=140,148,150,151) | 0 | 0 | 0 | 0
  Injection site Erythema (N=140,148,150,151) | 2 | 2 | 3 | 1
  Grade 3 Inj. site Erythema (N=140,148,150,151) | 0 | 0 | 0 | 0
  Injection-site Swelling (n=140,148,150,151) | 4 | 5 | 2 | 1
  Grade 3 Inj. site Swelling (n=140,148,150,151) | 0 | 2 | 0 | 0
  Injection site Induration (N=140,148,150,151) | 0 | 3 | 2 | 0
  Grade 3 Inj. site Induration (N=140,148,150,151) | 0 | 1 | 0 | 0
  Injection site Ecchymosis (N=140,148,150,151) | 1 | 0 | 2 | 1
  Grade 3 Inj. site Ecchymosis (N=140,148,150,151) | 0 | 0 | 0 | 0
  Fever (N=138,148,149,150) | 38 | 22 | 6 | 5
  Grade 3 Fever (N=138,148,149,150) | 1 | 0 | 0 | 0
  Headache (N=70,148,150,151) | 1 | 8 | 6 | 4
  Grade 3 Headache (N=70,148,150,151) | 0 | 0 | 0 | 0
  Malaise (N=70,148,150,151) | 5 | 11 | 6 | 5
  Grade 3 Malaise (N=70,148,150,151) | 1 | 0 | 0 | 0
  Myalgia (N=70,148,150,151) | 4 | 16 | 5 | 1
  Grade 3 Myalgia (N=70,148,150,151) | 0 | 0 | 0 | 0
  Shivering (N=70,148,150,151) | 1 | 6 | 3 | 0
  Grade 3 Shivering (N=70,148,150,151) | 0 | 0 | 0 | 0
  Crying abnormal (N=69,0,0,0) | 20 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Grade 3 Crying abnormal (N=69,0,0,0) | 0 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Drowsiness (N=69,0,0,0) | 12 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Grade 3 Drowsiness (N=69,0,0,0) | 1 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Appetite lost (N=69,0,0,0) | 20 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Grade 3 Appetite lost (N=69,0,0,0) | 4 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Irritability (N=69,0,0,0) | 14 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Grade 3 Irritability (N=69,0,0,0) | 0 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Vomiting (N=69,0,0,0) | 9 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group
  Grade 3 Vomiting (N =69,0,0,0) | 0 | NA — Event was not solicited in this group | NA — Event was not solicited in this group | NA — Event was not solicited in this group

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 56 post-vaccination.
Groups:
- Group 1: Participants 6 to 35 months of age received two 0.25 mL doses of trivalent influenza vaccine (split-virion, inactivated) given 28 days apart.
- Group 2: Participants 3 to 17 years of age received a single 0.5-mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Group 3: Participants 18 to 60 years of age received a single 0.5-mL dose of trivalent influenza vaccine (split-virion, inactivated).
- Group 4: Participants ≥61 years of age received a single 0.5-mL dose of trivalent influenza vaccine (split-virion, inactivated).
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 1/150 | 1/150 | 0/151 | 1/151
Other Adverse Events (participants affected / at risk) | 38/150 | 52/150 | 25/151 | 12/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=150) | Group 2 (N=150) | Group 3 (N=151) | Group 4 (N=151)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand foot and mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1 (N=150) | Group 2 (N=150) | Group 3 (N=151) | Group 4 (N=151)
Upper respiratory tract infection (Infections and infestations) | 21 (21) | 3 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 2 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 1 (1) | 0 (0) | 0 (0)
Injection site Pain/Tenderness (General disorders) | 38/140 (38) | 52/148 (52) | 25/150 (25) | 12 (12)
Fever (General disorders) | 38/138 (38) | 22/148 (22) | 6/149 (6) | 5/150 (5)
Headache (Nervous system disorders) | 1/70 (1) | 8/148 (8) | 6/150 (6) | 4 (4)
Malaise (General disorders) | 5/70 (5) | 11/148 (11) | 6/150 (6) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4/70 (4) | 16/148 (16) | 5/150 (5) | 1 (1)
Crying abnormal (Psychiatric disorders) | 20/69 (20) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Drowsiness (Nervous system disorders) | 12/69 (12) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Appetite lost (Metabolism and nutrition disorders) | 20/69 (20) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Irritability (Psychiatric disorders) | 14/69 (14) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Vomiting (Gastrointestinal disorders) | 9/69 (9) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Nasopharyngitis (Infections and infestations) | 10 (11) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications